CLINICAL TRIAL: NCT00885742
Title: A Prospective, Multicenter, Open-label, Phase 3b Study of Human Plasma-Derived Factor XIII Concentrate in Subjects With Congenital Factor XIII Deficiency
Brief Title: A Study of Factor XIII Concentrate in Subjects With Congenital Factor XIII Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BI71023_3001; 1482 (Other: CSL Behring); 2009-010722-19 (EudraCT Number)
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-06

CONDITIONS: Factor XIII Deficiency
Keywords: Hereditary Factor XIII deficiency; Factor XIII
MeSH Terms: conditions — Factor XIII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FXIII (Experimental): All subjects who received a dose of Factor XIII (FXIII) Concentrate (Human).
  Interventions: Biological: FXIII Concentrate (Human)

INTERVENTIONS:
Biological: FXIII Concentrate (Human) — Doses will be guided by the individual subject's most recent FXIII activity levels, with the objective of dosing every 28 days to maintain a trough FXIII activity level of approximately 5 to 20%.
  Subjects enrolled in this study who did not complete the pharmacokinetic study (Factor XIII Study BI71023_2002 [NCT00883090]) will initially receive FXIII Concentrate (Human) at a dose of 40 U/kg by intravenous (IV) infusion.
  Other Names: Fibrogammin-P

SUMMARY:
Congenital deficiency of factor XIII (FXIII) is an extremely rare inherited disorder associated with potentially life-threatening bleeding. Factor XIII Concentrate is given to patients whose blood is lacking factor XIII. Factor XIII Concentrate works by assisting blood in the usual clotting process, thereby preventing bleeding.

In this study, patients will be treated with FXIII Concentrate (Human) and followed closely to determine that they receive the dose that will best minimize the chance of bruising and bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent for study participation obtained before undergoing any study-specific procedures
* Documented congenital FXIII deficiency which requires prophylactic treatment with a FXIII containing product.
* Males and females of any age with congenital FXIII deficiency
* Received full hepatitis B vaccination and/or is hepatitis B surface antibody positive

Exclusion Criteria:

* Diagnosis of acquired FXIII deficiency
* Administration of a FXIII-containing product, including blood transfusions or other blood products within 4 weeks prior to the planned Day 0
* Any known congenital or acquired coagulation disorder other than congenital FXIII deficiency
* Known or suspected to have antibodies towards FXIII
* Use of any other investigational medicinal product within 4 weeks prior to the Baseline Visit (Day 0)
* Known Positivity for human immunodeficiency virus (HIV) or a positive result for HIV at the Screening Visit of this study or the FXIII study 2002 (NCT00883090).
* Serum aspartate transaminase (AST) or serum alanine transaminase (ALT) concentration >2.5 times the upper limit of normal at the Screening Visit of this study or at the Day 56 Visit of Factor XIII Study BI71023_2002 (NCT00883090)
* Fibrinogen level less than 85% of the lower limit of normal at the Screening Visit of this study or the Factor XIII Study BI71023_2002 (NCT00883090)
* Active bleeding ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 and/or ≥ moderate between the Screening and Baseline Visits
* Pregnant or breast-feeding
* Intention to become pregnant during the course of the study
* Female subjects of childbearing potential not using, or not willing to use, a medically reliable method of contraception for the entire duration of the study
* Suspected inability (e.g., language problems) or unwillingness to comply with study procedures or history of noncompliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (23):
- United States (22):
  - Study Site, Dothan, Alabama
  - Study Site, Oakland, California
  - Study Site, Orange, California
  - Study Site, San Francisco, California
  - Study Site, Stockton, California
  - Study Site, Hartford, Connecticut
  - Study Site, Fort Meyers, Florida
  - Study, Miami, Florida
  - Study Site, Boise, Idaho
  - Study Site, South Bend, Indiana
  - Study Site, Boston, Massachusetts
  - Study Site, Saint Paul, Minnesota
  - Study Site, Kansas City, Missouri
  - Study Site, Las Vegas, Nevada
  - Study Site, Lebanon, New Hampshire
  - Study Site, Newark, New Jersey
  - Study Site, Albany, New York
  - Study Site, New York, New York
  - Study Site, Chapel Hill, North Carolina
  - Study Site, Hershey, Pennsylvania
  - Study Site, Dallas, Texas
  - Study Site, Milwaukee, Wisconsin
- Study Site, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Derived] Ashley C, Chang E, Davis J, Mangione A, Frame V, Nugent DJ. Efficacy and safety of prophylactic treatment with plasma-derived factor XIII concentrate (human) in patients with congenital factor XIII deficiency. Haemophilia. 2015 Jan;21(1):102-8. doi: 10.1111/hae.12524. Epub 2014 Nov 7. PMID 25377187
- See also: Factor XIII Study BI71023_2002 (NCT00883090) — http://www.clinicaltrials.gov/ct2/show/NCT00883090?term=FXIII&rank=2
- See also: Factor XIII Study BI71023_3002 (NCT00945906) — http://clinicaltrials.gov/ct2/show/NCT00945906

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FXIII
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FXIII
Number analyzed (Participants) | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 20.1 (11.20)
Age, Customized [Number; unit: participants]
  < 16 years | 18
  16 to < 65 years | 23
  ≥ 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Spontaneous Bleeding Events Requiring Treatment (Treatment is Defined as Administration of a FXIII-Containing Product to Treat the Bleeding Event)
Description: The number of subjects requiring treatment with a Factor XIII-containing product to treat a spontaneous bleeding event.
Time Frame: Up to week 52
Population: The Efficacy Population comprised all subjects who received a dose of FXIII Concentrate (Human) during the study and included those who were assessed for efficacy at Baseline and had at least 1 follow-up FXIII activity trough level.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 41
participants | 0

2. Secondary Outcome: Association of the Incidence of Spontaneous Bleeding Events Requiring Treatment and FXIII Activity Trough Levels
Description: P-value determined from Generalized Estimating Equation (GEE) model parameter estimates with bleeding as the response variable and FXIII activity trough level as the explanatory variable.
Time Frame: 12 months
Population: The analysis population comprised those subjects with spontaneous bleeding events requiring treatment with a FXIII-containing product. Note: no subjects had spontaneous bleeding events requiring treatment with a FXIII-containing product, so no subjects were analyzed.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 0

3. Secondary Outcome: Adverse Events
Description: Number of subjects with any treatment-emergent adverse event (AE), treatment-related AE or serious AE (SAE). Treatment related AEs are defined as AEs whose relationship to study treatment is related, or possibly related, and AEs with missing relationship.
Time Frame: 12 months
Population: The Safety Population comprised all subjects who received a dose of FXIII Concentrate (Human) during the study.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 41
participants
  Any treatment-emergent AEs | 33
  Any treatment-emergent and treatment-related AE | 3
  Any treatment-emergent SAE | 4

4. Secondary Outcome: Peak FXIII Concentration at Steady State
Time Frame: At 12, 24, 36 and 48 weeks: at 30 and 60 minutes after the end of the infusion.
Population: The Pharmacokinetic (PK) Population comprised all subjects who received a dose of FXIII Concentrate (Human) during the study and included those who completed the study (defined as having sufficient bioanalytical assessments to calculate reliable estimates of the PK parameters).
Measure: Mean (Standard Deviation); unit: Units/mL
Arm/Group | FXIII
Number analyzed (Participants) | 41
Units/mL
  Week 12 (n = 40) | 0.968 (0.2292)
  Week 24 (n = 40) | 1.045 (0.3825)
  Week 36 (n = 41) | 0.962 (0.2306)
  Week 48 (n = 40) | 0.983 (0.2633)

5. Secondary Outcome: Trough FXIII Concentration at Steady State
Time Frame: At 12, 24, 36 and 48 weeks: immediately before infusion.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units/mL
Arm/Group | FXIII
Number analyzed (Participants) | 41
Units/mL
  Week 12 (n = 40) | 0.132 (0.0305)
  Week 24 (n = 41) | 0.136 (0.0362)
  Week 36 (n = 41) | 0.130 (0.0254)
  Week 48 (n = 41) | 0.150 (0.1138)

6. Secondary Outcome: Time to Peak Concentration
Time Frame: At 12, 24, 36 and 48 weeks: immediately before infusion, then at 30 and 60 minutes after the end of the infusion.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | FXIII
Number analyzed (Participants) | 41
Hour
  Week 12 (n = 40) | 0.632 (0.2296)
  Week 24 (n = 40) | 0.615 (0.1978)
  Week 36 (n = 39) | 0.623 (0.2350)
  Week 48 (n = 40) | 0.636 (0.2328)

7. Secondary Outcome: Incremental Recovery
Description: Incremental recovery (U/mL/U/kg) is defined as maximum (peak) FXIII activity (U/mL) obtained after infusion, per dose of (U/kg) infusion.
Time Frame: At 12, 24, 36 and 48 weeks: immediately before infusion, then at 30 and 60 minutes after the end of the infusion.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units/mL/Units/kg
Arm/Group | FXIII
Number analyzed (Participants) | 41
Units/mL/Units/kg
  Week 12 (n = 39) | 0.021 (0.0059)
  Week 24 (n = 38) | 0.023 (0.0104)
  Week 36 (n = 39) | 0.021 (0.0056)
  Week 48 (n = 38) | 0.020 (0.0056)

8. Secondary Outcome: Achievement of Trough Factor XIII Levels of 5% or Higher.
Description: Number of subjects with Factor XIII level ≥ 5% before infusion at Week 12, Week 24, Week 36 and Week 48.
Time Frame: At 12, 24, 36 and 48 weeks: immediately before infusion.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 41
participants
  Week 12 (n = 40) | 40
  Week 24 (n = 41) | 41
  Week 36 (n = 41) | 41
  Week 48 (n = 41) | 40

ADVERSE EVENTS:
Time Frame: 12 months
Description: The Safety Population comprised all subjects who received a dose of FXIII Concentrate (Human) during the study. Data presented for other, non-serious AEs are for treatment-emergent AEs.
Arm/Group | FXIII
Serious Adverse Events (participants affected / at risk) | 4/41
Other Adverse Events (participants affected / at risk) | 27/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FXIII (N=41)
Appendicitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hip injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic chest injury NOS (Injury, poisoning and procedural complications) | 1 (1)
Chest pain with radiation to left arm (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FXIII (N=41)
Vomiting (Gastrointestinal disorders) | 3 (6)
Fever (General disorders) | 5 (5)
Abrasions (Injury, poisoning and procedural complications) | 3 (5)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Bruising of thigh (Injury, poisoning and procedural complications) | 3 (3)
Thrombin-antithrombin III complex increased (Investigations) | 3 (5)
Wrist pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Upper respiratory infection (Infections and infestations) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to public release. The sponsor may request any changes necessary to prevent forfeiture of patent rights to data not in the public domain. For a multi-center study, the investigator must wait (i) at least 1 year after the study is completed at all sites or (ii) until notified by the sponsor that no multi-center publication is planned, before seeking publication review.